CLINICAL TRIAL: NCT04776668
Title: Living With Marfan Syndrome I: the Psychosocial and Health-related Quality of Life Effects of the Diagnosis for Aorto-vascular Manifestations (LIMA I Study)
Brief Title: Living With Marfan Syndrome and Your Aorta
Acronym: LIMA I
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Aortic Dissection Awareness UK & Ireland. (Other)
Responsible Party: Sponsor
Other Study IDs: 286206
Record Dates: First submitted 2021-02-18; First posted 2021-03-02 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Marfan Syndrome; Marfan Syndrome Cardiovascular Manifestations
MeSH Terms: conditions — Marfan Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Marfan Syndrome (MFS) is a genetic disease affecting the eyes, skeleton, heart and arteries. Despite MFS affecting multiple organ systems, cardiovascular manifestations are the most serious and life threatening. Approximately 80% of adult MFS patients will have a dilated aortic root by age 40 years with aortic aneurysm and dissection the leading causes of morbidity and mortality. Thus, MFS patients require lifelong cardiac surveillance. Living with a diagnosis of Marfan Syndrome and aorto-vascular manifestations affects patients' mental health, well-being and quality of life in ways that are not well understood.

This study will address the current knowledge gaps in this area and will provide the information needed to design interventions for MFS patients with aorto-vascular problems to help improve the patients' mental health, well-being and quality of life. The study will include adult MFS patients who have been diagnosed with aorto-vascular problems.

The overall aim of the study is to explore the psychosocial and health-related quality of life (HRQoL) effects of the diagnosis for aorto-vascular manifestations of MFS in 3 large UK cardiac centres. To achieve this, the researchers will ask the potential participants, after obtaining informed consent, to complete a series of accepted/validated questionnaires to measure the study participants' health-related quality of life (SF-36 and EQ5D questionnaire) and psychosocial factors such as depression (CES-D questionnaire), fatigue (Fatigue Severity Scale), stigma (Perceived Stigma Questionnaire), self-esteem (Rosenberg Self-esteem Scale), pain and illness perception (Illness Perception Questionnaire). The researcher will also conduct a one-to-one semi-structured interview with some participants to identify factors important to patients that are not captured in the questionnaires used.

DETAILED DESCRIPTION:
Marfan Syndrome (MFS) is a rare autosomal-dominant connective tissue disorder with pleiotropic manifestations primarily affecting the skeletal, ocular, and cardiovascular systems. Despite MFS affecting multiple organ systems, cardiovascular manifestations are the most serious and life threatening. Approximately 80% of adult MFS patients will have a dilated aortic root by age 40 years with aortic aneurysm and dissection the leading causes of morbidity and mortality, requiring lifelong cardiac surveillance. Since diagnosis is made on average at 19 years old and life expectancy has increased considerably from 32 years in the 1970s, to 41 years in the 1990s and is now comparable to the general population (with the introduction of prophylactic aortic surgery), MFS patients have to live knowing that at least one major heart surgery is required in the patients' lifetime. Further, from the researchers' clinical experience, not all individuals with MFS perceived their cardiovascular conditions as treatable. Hence, the impact of knowing that they have aortovascular manifestations may be more striking than in other age and sex-matched cardiac surgical population. To date, there is still no available study assessing the impact of this diagnosis on the health-related quality of life (HRQoL) and psychosocial aspect of MFS patients.

The overarching aim of the study is to explore the psychosocial and HRQoL effects of the diagnosis for aorto-vascular manifestations of MFS in three large UK cardiac centres. This will be achieved using a mixed-method approach consisting of two studies. Study 1 (S1) is a quantitative observational exploratory study while Study 2 (S2) is a qualitative exploratory study using semi-structured interviews to identify factors important to patients that are not captured in the questionnaires used in S1. Potential participants will be recruited from the aortopathy clinic. HRQoL and psychosocial factors will be determined and quantified using validated questionnaires which will be delivered either in paper or electronic format, depending on participants' preference.

The outcome of the study will contribute to the UK and international evidence-base on the HRQoL and psychosocial impact of the diagnosis of aortovascular manifestations on MFS patients. The result will also be useful to better understand the condition and potentially guide the researchers in devising a patient care pathway that includes this aspect of care as well as develop a holistic and comprehensive service for this patient group.

ELIGIBILITY:
Inclusion Criteria:

1. >/= 18 years old;
2. have validated diagnosis of MFS (using revised Ghent criteria);
3. diagnosed with aorto-vascular manifestations

Exclusion Criteria:

1. <18years old
2. Unable or unwilling to give written informed consent.
3. Inability to understand written and/or verbal English

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible consecutive patients with a diagnosis of MFS at three large UK cardiac centres will be identified from the aortopathy clinic by a member of the cardiac clinical care team.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Health-related Quality of Life (HRQoL) | 24 hours after consent is obtained
  HRQoL will be measured using the Short Form Health Survey 36 (SF-36). SF-36 consists of 8 sub-scales. All scales do contribute in different proportions to the scoring of the physical and mental dimensions, represented by the Physical Component Summary (PCS) and Mental Component Summary (MCS). Using an algorithm, raw scores can be converted to a transformed scale scores ranging from 0-100, with higher score indicating a better health state.
Health-related Quality of Life (HRQoL) | 24 hours after consent is obtained
  HRQoL will be measured using EQ-5D. EQ-5D is divided into 2 components: health care description and evaluation. In the description part, summation of score ranges from 1 to 3; with 1 indicates the best health state and 3 indicates more severe or frequent problem. The evaluation part utilises a visual analogue scale to indicate the general health status with 100 indicating the best health status and 0 indicating the worst health status.

SECONDARY OUTCOMES:
Psychosocial factor: depression | 24 hours after consent is obtained
  Depression will be measured using Centre for Epidemiological Studies Depression Scale (CES-D). The overall score ranges from 0 to 60, with higher scores indicating a more severe depressive symptoms. In general population, a cut-off score of 16 or above is used to identify those with significant clinical signs of depression.
Psychosocial factor: fatigue | 24 hours after consent is obtained
  Fatigue will be determined using Fatigue Severity Scale (FSS). The minimum possible score is 9 and maximum possible score is 63. Higher score indicates greater fatigue severity.
Psychosocial factor: stigma | 24 hours after consent is obtained
  Stigma will be measured using Perceived Stigma Questionnaire (PSQ). PSQ is composed of 4 sub-scales. Score on each sub-scale ranges from 1 to 6. Mean scores of >/= 2.0 on the devaluation and discrimination sub-scale indicates feeling of discriminated against or devalued. Mean scores of </= 3.5 on the withdrawal and secrecy sub-scales and </= 2.0 on the education sub-scale indicates the use of secrecy / withdrawal and education as coping styles, respectively.
Psychosocial factor: self esteem | 24 hours after consent is obtained
  Self-esteem will be measured using Rosenberg Self-esteem Scale (RSS); score ranges from 10 (min) -40 (max); higher score indicates higher self-esteem.
Psychosocial factors: pain and illness perception | 24 hours after consent is obtained
  Pain and Illness Perception will be determined using Illness Perception Questionnaire (IPQ). IPQ is divided into 5 components. The identity component is scored by summing the number of items identified at 'occasionally' or greater resulting to a total score ranging from 0 to 12 for the core list. The four other components are presented in mixed order and can be rated using a 5-point Likert scale ranging from 'strongly disagree' (1) to 'strongly agree (5).

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomews Hospital, London, United Kingdom